CLINICAL TRIAL: NCT03310853
Title: The Effect of Probiotics on Maintenance of Health in Pregnancy and Infants: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: The Effect of Probiotics on Maintenance of Health in Pregnancy and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MOM study
Record Dates: First submitted 2017-09-28; First posted 2017-10-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy
Keywords: probiotics; infections; bacterial vaginosis
MeSH Terms: conditions — Infections; Vaginosis, Bacterial | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Combination of two probiotic strains in one capsule
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Non active ingredients in a capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dosing regimen of one capsule daily for a maximum of 18 weeks
  Arms: Probiotic
Other: Placebo — Dosing regimen of one capsule daily for a maximum of 18 weeks
  Arms: Placebo

SUMMARY:
This phase 2 study evaluates the effect of perinatal use of probiotics on the number of diagnosed viral, bacterial and fungal infections in pregnant women and on the maintenance of a health pregnancy. In addition, the effect of probiotics intake during pregnancy and breastfeeding on the infant's overall health status will be evaluated.

DETAILED DESCRIPTION:
Throughout pregnancy women undergo many biological changes, including alterations in their microbiota. These infections can exacerbate pregnancy complications and increase the risk of preeclampsia and preterm birth. The present study aims to evaluate the potential effects of perinatal use of probiotics on the number of diagnosed viral, bacterial and fungal infections in pregnant women and on the maintenance of a healthy pregnancy. Potential infections include but are not limited to influenza/colds, bacterial vaginosis, mastitis, candidiasis, urinary tract infection and gingivitis. Additionally, the benefits of probiotic intake by the mother on the infant during pregnancy and breastfeeding will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Less than 28 weeks of gestation (3rd trimester)
* ≥18 to <40 years old
* Singleton gestation
* Availability and willingness to come in for morning visits
* Planning to breastfeed
* Willing to complete questionnaires, records, and diaries associated with the study and to complete all clinical visits
* Willing to discontinue consumption of fermented foods (e.g. foods that contain probiotics such as Kefir, pickles, etc.) or probiotics (e.g. yogurts with live active cultures or probiotic supplements)
* Able to provide informed consent

Exclusion Criteria:

* Known gestational diabetes or diabetes type 1 or 2
* Known blood/bleeding disorders
* Known liver and kidney disorders
* Known unstable cardiovascular diseases
* Women with a personal history of or currently diagnosed with preeclampsia
* Suffering from neurological diseases (e.g. Alzheimer's disease, Parkinson's disease, epilepsy, etc.)
* Suffering from gastrointestinal diseases (e.g. gastric ulcers, Crohn's disease, ulcerative colitis, etc.)
* Current symptoms of depression or experienced depressive symptoms in the past 2 years
* Maternal history of second trimester loss
* Women diagnosed HIV Positive or with Hepatitis B or C
* Known fetal abnormality
* Daily use of probiotic product within 2 weeks of the screening visit. The potential participant could be eligible to participate after a 2-week wash-out period
* Use of any antibiotic drug within 1 month of screening. The potential participant could be eligible to participate after a 2-week wash-out period
* Smoking, alcohol consumption or drug use during pregnancy
* History of alcohol or substance abuse six months prior to screening
* Allergies to milk, soy, or yeast

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Number of diagnosed infections in pregnant women | up to 12 weeks
  This includes any viral, bacterial and fungal infection (e.g. bacterial vaginosis, candidiasis, urinary tract infection, mastitis, cold, flu, gingivitis, etc.). A vaginal swab and saliva sample will be taken at every visit on site throughout pregnancy. The vaginal swab will be used for the detection of Bacterial Vaginosis and Candidiasis. Other required swab samples will be collected if an infection occurs (e.g. vaginal, mouth, throat, nose, etc.). If an infection is suspected by a participant in-between a scheduled visit, the participant will come on site to be checked by a doctor. If the participant is subsequently diagnosed with an infection, a saliva sample will need to be taken at this time.

SECONDARY OUTCOMES:
Levels of glucose, insulin, triglycerides and iron | Measured 2 times up to 12 weeks
  Assessed via blood sample throughout the pregnancy
Vaginal mycobiota | Measured 3 times up to 18 weeks
  Vaginal microbiome which includes bacteria, fungus and potentially other eukaryotic micro-organisms such as parasites or viruses. To be assessed with a vaginal swab during pregnancy and after delivery.
Inflammatory markers | Measured up to 3 times in the 18 week time frame
  Assessing levels of both pro- and anti- inflammatory markers in the mother during pregnancy (through stool and blood samples) and after delivery (through breast milk sample).
Vaginal microbiota | Measured 3 times up to 18 weeks
  Effects of the probiotic interventions on overall microbiota composition in the mother will be assessed. In addition, recovery of the probiotic strains in the vaginal samples will be assessed.
Premature rupture of membranes (PROM) | Measured 1 time at week 12
  Incidence of PROM on the probiotic versus the group
Levels of secretory immunoglobulin A (sIgA) in the mother | Measured up to 4 times in the 18 week time frame
  Assessed via saliva samples throughout pregnancy and a breast milk sample after delivery.
Levels of secretory immunoglobulin A (sIgA) in the infant | Measured 1 time up to18 weeks
  Assessed via stool sample after birth.
Gut microbiota in the mother | Measured 3 times up to 18 weeks
  Effects of the probiotic interventions on overall microbiota composition will be assessed. In addition, recovery of the probiotic strains in the stool samples will be assessed.
Gut microbiota in the infant | Measured 1 time up to 18 weeks
  Effects of the probiotic interventions on overall microbiota composition will be assessed. In addition, recovery of the probiotic strains in the stool samples will be assessed.
Stool frequency and consistency in the mother | Self-reported, daily up to 18 weeks
  Assessed with the Bristol Stool Scale
Stool frequency and pattern in the infant | Self-reported by the mother, daily up to 4-6 weeks
  Assessed with the Amsterdam Infant Stool Scale
Weight in the mother | Measured 3 times up to 18 weeks. Pre-pregnancy weight will also be noted via information collection on a demographic questionnaire.
  To assess change in body weight
Breast milk microbiota | Measured 1 time up to 18 weeks
  Effects of the probiotic interventions on overall microbiota composition will be assessed. In addition, recovery of the probiotic strains in the breast milk samples will be assessed.
Post-Partum Depression | Measured 2 time up to 18 weeks
  To be assessed with the Edinburgh Postnatal Depression Scale
Infant's health status - NEC | Measured 1 time up to 18 weeks.
  To assess the probability of an infant with NEC
Anthropometric measurements | Measured 1 time up to 18 weeks. The infant's anthropometric measurements at birth will also be noted.
  Crown-heel length and head circumference
Weight in the infant | Measured 2 times up to 18 weeks.
  To assess change in body weight
Crying time in the infant | Self-reported by the mother, daily up to 4-6 weeks
  To assess the mean daily crying time of infants
Colic in the infant | Self-reported by the mother, daily up to 4-6 weeks
  To asses the probability of an infant with colic
Sleep in the infant | Self-reported by the mother, daily up to 4-6 weeks
  Number of total hours and number of consecutive hours
Number of infections | Self-reported by the mother, daily up to 4-6 weeks
  To assess the number of infections
Skin diseases or conditions | 1 year follow up phone call
  Skin diseases/conditions as well as the child's overall health status 1 year after birth will be assessed.
Infant's health status - jaundice | Measured 1 time up to 18 weeks.
  To assess the probability of an infant with jaundice
Infant's health status - Hyperbilirubinemia | Measured 1 time up to 18 weeks.
  To assess the probability of an infant with Hyperbilirubinemia

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique OVO, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No